CLINICAL TRIAL: NCT02969980
Title: Allogeneic Hematopoietic Cell Transplantation Using Post-transplantation Cyclophosphamide in Myelodysplastic Syndrome Patients
Brief Title: Hematopoietic Cell Transplantation With Post-transplantation Cyclophosphamide in MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, M.D. Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS_PTCy_2016
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; AML progressed from MDS; CMML
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Cyclophosphamide

ARMS (1):
- PTCy (Experimental): Patients who receive post-transplantation cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/kg/day i.v. daily on days 3 and 4 of hematopoietic cell transplantation

SUMMARY:
This study is conducted to evaluate the feasibility and efficacy of post-transplantation cyclophosphamide with myeloablative or reduced-intensity conditioning regimen for allogeneic hematopoietic cell transplantation (HCT) in patients with myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
* Conditioning regimen A) Busulfan 3.2 mg/kg/day i.v. daily For 4 days (days -7 to -4) in patients aged < 55 years For 2 days (days -7 and -6) in patients aged ≥ 55 years B) Fludarabine 30 mg/m2/day i.v. daily on days -7 to -2 (for 6 days)
* Harvest and infusion of donor hematopoietic cells Harvested peripheral blood mononuclear cells of donors via leukapheresis will be infused to recipients on day 0. Additional infusion on day 1 can be made based on the judgement of attending physician.
* GVHD prophylaxis A) Cyclophosphamide 50 mg/kg/day i.v. daily on days 3 and 4 (for 2 days) B) Cyclosporine: 1.5 mg/kg i.v. every 12 h hours beginning on day 5 and changed to oral dosing when oral intake is possible. If there is no evidence of GVHD, the dosage will be tapered beginning on day 90 and discontinued on day 180. C) MMF: 15 mg/kg p.o. 3 times daily with a maximum daily dose of 3.0 g beginning on day 5

If there is no active GVHD, Cyclosporine and MMF will be discontinued without taper at day 180 and 35, respectively.

ELIGIBILITY:
Inclusion Criteria:

* MDS defined by WHO classification, chronic myelomonocytic leukemia (CMML), or acute myeloid leukemia (AML) evolving from MDS A. IPSS > 1.0 or bone marrow blast ≥ 5% at any time points before HCT or B. AML progressed from MDS or C. CMML
* Patients receiving first HCT
* Patients with appropriate hematopoietic cell donors A. HLA-matched sibling donor B. Unrelated donor C. HLA-mismatched familial donor
* 15 years old or older
* Adequate performance status (Karnofsky score of 70 or more)
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 3.0 x upper normal limit, and creatinine < 2.0 mg/dL).
* Adequate cardiac function (left ventricular ejection fraction over 40% on heart scan or echocardiogram
* Signed and dated informed consent must be obtained from both recipient and donor.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
the incidence of acute and chronic graft-versus-host disease | 100 days and 2 year, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea